CLINICAL TRIAL: NCT03570931
Title: A Prospective Open-label Study to Assess Efficacy and Safety of RT001 in Subjects With Infantile Neuroaxonal Dystrophy
Brief Title: A Study to Assess Efficacy and Safety of RT001 in Subjects With Infantile Neuroaxonal Dystrophy
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biojiva LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT001-008
Record Dates: First submitted 2018-06-11; First posted 2018-06-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Infantile Neuroaxonal Dystrophy
Keywords: INAD; Infantile Neuroaxonal Dystrophy
MeSH Terms: conditions — Neuroaxonal Dystrophies | interventions — RT001

STUDY DESIGN:
Intervention Model Description: Single arm open-label study
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RT001 (Experimental): RT001, oral, 3.84 g/day
  Interventions: Drug: RT001

INTERVENTIONS:
Drug: RT001 — RT001 is encapsulated di-deutero synthetic homologue of linoleic acid ethyl ester. Each capsule contains 960 mg of RT001.
  Other Names: Deuterated linoleic acid

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of RT001 in patients with Infantile Neuroaxonal Dystrophy (INAD).

DETAILED DESCRIPTION:
This is a single arm open-label study with a structured observation of INAD patients treated with RT001. Enrolled subjects will undergo observation and testing to determine the effect of RT001 treatment. Fifteen to twenty eligible subjects will be treated with RT001 for long-term evaluation of efficacy, safety, tolerability, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 months to 10 years of age
2. Medical history consistent with the symptoms of classic INAD (onset of symptoms between the ages of 6 months and 3 years)
3. Homozygous for PLA2G6 deficiency (variant alleles may be mixed heterozygotes)
4. Must have impairment in at least 2 of the assessed categories at baseline
5. Signed informed consent form (ICF) prior to entry into the study
6. Able to provide the necessary blood samples

Exclusion Criteria:

1. Received treatment with other experimental therapies within the last 30 days prior to the first dose
2. Requiring mechanical ventilation, other than positive air pressure support primarily for mitigation of sleep apnea.
3. Have a life expectancy of less than one year
4. Diagnosis of atypical NAD (ANAD)
5. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to return for visits as scheduled

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Spasticity Scale | 12 months
  Change from baseline in the Modified Ashworth spasticity scale.

SECONDARY OUTCOMES:
INAD Progression Composite | 12 months
  Change from baseline in an INAD composite score to assess the overall treatment effect on the most progressive aspects of the disease
Progression Free Survival Time | All available data
  Progression free survival time (mortality or pneumonia)

OTHER OUTCOMES:
Modified Infantile Neuroaxonal Dystrophy Rating Scale (mINAD-RS24) | 12 months
  Change in score from baseline derived from a structured pediatric neurological development exam tailored for INAD, involving elements of activities of daily living and vital functions.
Modified Parental Rating Scale (mPRS22) | 12 months
  Change in score from baseline from a parental rating scale tailored for INAD, involving elements of activities of daily living and vital functions
Original Infantile Neuroaxonal Dystrophy Rating Scale (INAD-RS40) | 12 months
  Change in score from baseline derived from a structured pediatric neurological development exam tailored for INAD, involving elements of activities of daily living and vital functions.
Original Parental Rating Scale (mPRS33) | 12 months
  Change in score from baseline from a parental rating scale tailored for INAD, involving elements of activities of daily living and vital functions
Incidence of Treatment-Emergent Adverse Events | 12 months
  The incidence of treatment-emergent adverse events will be presented by severity and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milner, MD, Study Director — Chief Medical Officer
Locations (2):
- United States (2):
  - University of California San Francisco, Benioff Children's Hospital, San Francisco, California
  - Jacobs Levy Genomics and Research Program, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided